CLINICAL TRIAL: NCT03078751
Title: An Open Label, Multi-center Protocol for U.S. Patients Enrolled in a Study of Ribociclib With Endocrine Therapy as an Adjuvant Treatment in Patients With Hormone Receptor-positive, HER2-negative, High Risk Early Breast Cancer
Brief Title: Adjuvant Ribociclib With Endocrine Therapy in Hormone Receptor+/HER2- High Risk Early Breast Cancer
Acronym: EarLEE-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLEE011G2301; 2014-001795-53 (EudraCT Number)
Record Dates: First submitted 2017-02-27; First posted 2017-03-13 (Actual); Results first posted 2021-01-15 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer
Keywords: Hormone receptor-positive; Estrogen and/or progesterone receptor-positive; HER2-negative; High risk early breast cancer; Adjuvant; Ribociclib; LEE011; CDK4/6 inhibitor; Endocrine therapy; Phase II; Breast carcinoma; Breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib

STUDY DESIGN:
Masking Description: The trial used to be a placebo-controlled, blinded trial. It was amended to an open-label trial after protocol amendment 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ribociclib + adjuvant endocrine therapy (ET) (Experimental): Patients in this arm took Ribociclib in combination with standard adjuvant endocrine therapy.
  ET was one of these 4: Letrozole, Anastrozole, Exemestane, Tamoxifen (Tamoxifen no longer permitted after protocol amendment 2)
  Interventions: Drug: Ribociclib; Drug: Adjuvant endocrine therapy
- Placebo + adjuvant endocrine therapy (ET) (Placebo Comparator): Patients in this arm took Placebo in combination with standard adjuvant endocrine therapy. ET was one of these 4: Letrozole, Anastrozole, Exemestane, Tamoxifen
  Interventions: Drug: Adjuvant endocrine therapy; Drug: Placebo

INTERVENTIONS:
Drug: Ribociclib — Ribociclib 600 mg daily on days 1 to 21 of a 28-day cycle for 26 cycles (approximately 24 months).
  Ribociclib was supplied in the form of 200 mg film-coated tablets taken by mouth.
  Other Names: LEE011
  Arms: Ribociclib + adjuvant endocrine therapy (ET)
Drug: Adjuvant endocrine therapy — Letrozole 2.5 mg by mouth daily, or anastrozole 1 mg by mouth daily, exemestane 25 mg by mouth daily, tamoxifen 20 mg by mouth daily, for a total duration of at least 60 months. In premenopausal women, a GnRH agonist administered every 28 days.
Drug: Placebo — Placebo 600 mg daily on days 1 to 21 of a 28-day cycle for 26 cycles (approximately 24 months).
  Placebo was supplied in the form of 200 mg film-coated tablets taken by mouth.
  Arms: Placebo + adjuvant endocrine therapy (ET)

SUMMARY:
This was an open label, multi-center protocol for U.S. patients enrolled in the study of ribociclib with endocrine therapy as an adjuvant treatment in patients with hormone receptor-positive, HER2-negative, high risk early breast cancer

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the preliminary safety and tolerability of ribociclib to standard adjuvant endocrine therapy (ET) in patients with hormone receptor (HR) positive, Human Epidermal Growth Factor Receptor2 (HER2) negative high risk early breast cancer (EBC).

Originally, this was a randomized, Phase III, double-blind, placebo-controlled, multi-center, international study to evaluate efficacy and safety of ribociclib with ET as an adjuvant treatment in patients with HR-positive, HER2-negative, high risk EBC.

Patients were randomized at a ratio of 1:1 to receive either ribociclib or placebo for approximately 24 months in combination with a standard adjuvant ET with ET continued for at least 60 months.

However, following a review of the ribociclib development program strategy, a decision was taken to explore a different approach by initiating a single Phase III study for simplicity of trial logistics and for the purpose of analyzing the overall population through a single clinical trial. Therefore, this study was closed to enrollment early and was amended to be an open label, multi-center Phase II study conducted in the US only. All randomized patients were unblinded; patients randomized to placebo were permanently discontinued from the study and patients randomized to ribociclib were offered the option to continue treatment with ribociclib + ET.

The study included a screening phase (28 days), a treatment phase composed of maximum of 26 cycles of ribociclib in combination with ET (approximately 24 months) or until disease recurrence, intolerable toxicity, withdrawal of consent, or discontinuation from the study treatment for any other reason, whichever was earlier, and a 30 days safety follow up from last dose of ribociclib. Ribociclib was given orally once a day on days 1 to 21 in each 28 days cycle.

Safety was assessed for each patient until 30 days after the last dose of ribociclib and included routine safety monitoring except in case of death, loss to follow up or withdrawal of consent.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed unilateral primary invasive adenocarcinoma of the breast
* Estrogen receptor-positive and/or progesterone receptor-positive, HER2-negative breast cancer
* Patient is after surgical resection of the tumor where tumor was removed completely, with the final surgical specimen microscopic margins free from tumor and with available archival tumor tissue from the surgical specimen
* Patient who received adjuvant chemotherapy and have AJCC 8th edition Prognostic Stage Group III tumor; or patient who received neoadjuvant chemotherapy and have 1 or more ipsilateral axillary lymph nodes with residual tumor metastases greater than 2.0 mm in lymph node(-s) and residual tumor greater than 10.0 mm in breast tissue
* Patient has completed multi-agent adjuvant or neoadjuvant chemotherapy of ≥ 4 cycles or ≥ 12 weeks which included taxanes prior to screening
* Patient has completed adjuvant radiotherapy (if indicated) prior to screening
* Patient may already have initiated adjuvant endocrine therapy (ET) at the time of randomization, but randomization must take place within 52 weeks of date of initial histological diagnosis of breast cancer and within 12 weeks of initiating ET
* ECOG Performance Status 0 or 1
* Adequate bone marrow and organ function
* Sodium, potassium, phosphorus, magnesium and total calcium laboratory values within normal limits
* QTcF interval < 450 msec and mean resting heart rate 50-90 bpm

Key Exclusion Criteria:

* Prior treatment with CDK4/6 inhibitor
* Prior treatment with tamoxifen, raloxifen or aromatase inhibitors for reduction in risk (chemoprevention) of breast cancer and/or treatment for osteoporosis within last 2 years
* Prior treatment with anthracyclines at cumulative doses of 450 mg/m² or more for doxorubicin or 900 mg/m² or more for epirubicin
* Distant metastases of breast cancer beyond regional lymph nodes
* Patient has not recovered from clinical and laboratory acute toxicities of chemotherapy, radiotherapy and surgery
* Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality, or clinically significant cardiac arrhythmias
* Uncontrolled hypertension with systolic blood pressure >160 mmHg
* Patient is currently receiving any of the prohibited substances that cannot be discontinued 7 days prior to Cycle 1 Day 1: concomitant medications, herbal supplements, and/or fruits and their juices that are known as strong inhibitors or inducers of CYP3A4/5; medications that have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5; systemic corticosteroids ≤ 2 weeks prior to starting study drug, or who have not fully recovered from side effects of such treatment; concomitant medications with a known risk to prolong the QT interval and/or known to cause torsades de points that cannot be discontinued or replaced by safe alternative medication.
* Pregnant or breast-feeding (lactating) women or women who plan to become pregnant or breast-feed during the study
* Women of child-bearing potential unless they are using highly effective methods of contraception during the study treatment and for 21 days after stopping the study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (33):
- United States (33):
  - Arizona Oncology Associates PC- HAL, Tucson, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
  - CBCC Global Research, Bakersfield, California
  - University of California - Los Angeles, Los Angeles, California
  - Ventura County Hematology and Oncology, Oxnard, California
  - TRIO - Torrance Health Association, Redondo Beach, California
  - Innovative Clinical Research Institute, Whittier, California
  - Rocky Mountain Cancer Centers Regulatory, Denver, Colorado
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Florida Cancer Specialists South Region, Fort Myers, Florida
  - Memorial Regional Hospital, Hollywood, Florida
  - Hematology Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - Florida Cancer Specialists - North Florida Cancer Specialist N, St. Petersburg, Florida
  - Northside Hospital Central Research Dept., Atlanta, Georgia
  - Summit Cancer Care, PC, Savannah, Georgia
  - Health Midwest Ventures Group, Inc d/b/a HCA MidAmerica Div., Leawood, Kansas
  - Maryland Oncology Hematology P A, Silver Spring, Maryland
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Barnabas Medical Center 2nd Floor East Wing, Livingston, New Jersey
  - Pro Health Care Associates, New Hyde Park, New York
  - The Presbyterian Hospital, Charlotte, North Carolina
  - Tennessee Oncology, PLLC, Chattanooga, Tennessee
  - The West Clinic, Germantown, Tennessee
  - SCRI - Tennessee Oncology, Nashville, Tennessee
  - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology P A Texas Oncology - Houston, Dallas, Texas
  - Millennium Oncology, Houston, Texas
  - Cancer Care Network of South Texas, San Antonio, Texas
  - Texas Oncology PA - Tyler, Tyler, Texas
  - Fairfax Northern Virginia Hem/Onc, Fairfax, Virginia
  - Multicare Institute for Research and Innovation, Tacoma, Washington
  - Northwest Medical Specialties, Tacoma, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the triasl in line with applicable laws and regulations.
  This trial data will be available according to the process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Result] Hudis CA, Barlow WE, Costantino JP, Gray RJ, Pritchard KI, Chapman JA, Sparano JA, Hunsberger S, Enos RA, Gelber RD, Zujewski JA. Proposal for standardized definitions for efficacy end points in adjuvant breast cancer trials: the STEEP system. J Clin Oncol. 2007 May 20;25(15):2127-32. doi: 10.1200/JCO.2006.10.3523. PMID 17513820
- [Result] Hortobagyi GN, Connolly JL, D'Orsi CJ, et al (2017). Breast. From AJCC Cancer Staging Manual 8th ed. By Amin MB, Edge S, Greene FL, et al. Springer
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=724

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was closed early for recruitment and amended into an open-label, multi-centre, Phase II, conducted in the US only. A total of 54 patients were enrolled and randomized (26 in the ribociclib + ET arm and 28 in placebo + ET arm) at the time of recruitment closure. All randomized patients were unblinded. Patients randomized to placebo were permanently discontinued from the study and patients on ribociclib + ET were offered the option to continue treatment.
Pre-assignment Details: Approximately 2000 patients were planned to be enrolled in the study.
Period: Overall Study
Arm/Group | Ribociclib + Adjuvant Endocrine Therapy (ET) | Placebo + Adjuvant Endocrine Therapy (ET)
Started | 26 | 28
Untreated Participants | 0 | 4
Safety Set | 26 | 24
Completed | 13 | 0
Not Completed | 13 | 28
Not completed — Adverse Event | 4 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Terminated by Sponsor = early terminated recruitment | 0 | 23
Not completed — Subject/guardian decision | 8 | 1
Not completed — Untreated | 0 | 4

BASELINE CHARACTERISTICS:
Population: Full Analysis set (FAS) includes all randomized patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Ribociclib + Adjuvant Endocrine Therapy (ET) | Placebo + Adjuvant Endocrine Therapy (ET) | Total
Number analyzed (Participants) | 26 | 28 | 54
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.7 (11.23) | 54.7 (9.04) | 55.7 (10.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 28 | 54
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 2 | 3 | 5
  Black | 3 | 4 | 7
  Caucasian | 18 | 19 | 37
  Other | 2 | 1 | 3
  Unknown | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: These are the number of participants who had adverse events or serious adverse events regardless of whether is was suspected to be drug-related or not
Time Frame: Up to 26 months
Population: Safety set includes all patients who received at least one dose of any component of study treatment
Measure: Number; unit: Participants
Arm/Group | Ribociclib + Adjuvant Endocrine Therapy (ET) | Placebo + Adjuvant Endocrine Therapy (ET)
Number analyzed (Participants) | 26 | 24
Participants
  Adverse Events | 25 | 21
  Serious Adverse Events | 4 | 2

2. Primary Outcome: Percentage of Participants With Adverse Events and Serious Adverse Events
Description: These are the percentage of participants that had adverse events or serious adverse events regardless of whether is was suspected to be drug-related or not
Time Frame: Up to 26 months
Population: Safety set includes all patients who received at least one dose of any component of study treatment
Measure: Number; unit: Percentage of participants
Arm/Group | Ribociclib + Adjuvant Endocrine Therapy (ET) | Placebo + Adjuvant Endocrine Therapy (ET)
Number analyzed (Participants) | 26 | 24
Percentage of participants
  Adverse Events | 96.2 | 87.5
  Serious Adverse Events | 15.4 | 8.3

ADVERSE EVENTS:
Time Frame: Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 28 days post treatment, up to maximum duration of approx. 26 months
Description: Any sign or symptom that occurs during the study treatment plus 28 days post treatment.
Arm/Group | Ribociclib + Adjuvant Endocrine Therapy (ET) | Placebo + Adjuvant Endocrine Therapy (ET)
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 4/26 | 2/24
Other Adverse Events (participants affected / at risk) | 25/26 | 19/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ribociclib + Adjuvant Endocrine Therapy (ET) (N=26) | Placebo + Adjuvant Endocrine Therapy (ET) (N=24)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Breast cellulitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ribociclib + Adjuvant Endocrine Therapy (ET) (N=26) | Placebo + Adjuvant Endocrine Therapy (ET) (N=24)
Anaemia (Blood and lymphatic system disorders) | 6 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 14 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0
Palpitations (Cardiac disorders) | 2 | 0
Vision blurred (Eye disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 6 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 0
Nausea (Gastrointestinal disorders) | 12 | 6
Stomatitis (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 4 | 3
Axillary pain (General disorders) | 1 | 2
Chest pain (General disorders) | 2 | 0
Fatigue (General disorders) | 12 | 1
Influenza like illness (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 3 | 1
Pain (General disorders) | 3 | 0
Pyrexia (General disorders) | 4 | 1
Herpes zoster (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 2 | 2
Nasopharyngitis (Infections and infestations) | 5 | 0
Pneumonia (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 5 | 1
Urinary tract infection (Infections and infestations) | 3 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 1
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0
Alanine aminotransferase increased (Investigations) | 5 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 0
Blood calcium decreased (Investigations) | 2 | 0
Blood cholesterol increased (Investigations) | 2 | 0
Blood creatinine increased (Investigations) | 4 | 0
Lymphocyte count decreased (Investigations) | 4 | 0
Neutrophil count decreased (Investigations) | 7 | 0
Weight increased (Investigations) | 2 | 0
White blood cell count decreased (Investigations) | 10 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1
Dizziness (Nervous system disorders) | 4 | 2
Dysgeusia (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 5 | 2
Neuropathy peripheral (Nervous system disorders) | 2 | 0
Confusional state (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 2
Pollakiuria (Renal and urinary disorders) | 2 | 0
Breast pain (Reproductive system and breast disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Hot flush (Vascular disorders) | 3 | 3
Lymphoedema (Vascular disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study. Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed. The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/51/NCT03078751/Prot_001.pdf
  • Statistical Analysis Plan (2020-02-24): https://cdn.clinicaltrials.gov/large-docs/51/NCT03078751/SAP_000.pdf